CLINICAL TRIAL: NCT03052478
Title: Phase II, Single-arm Study of Vismodegib in Advanced Gastric Adenocarcinoma Patients With SMO Overexpression
Brief Title: Study of Vismodegib in Advanced Gastric Adenocarcinoma Patients With SMO Overexpression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeeyun Lee, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-08-130
Record Dates: First submitted 2017-02-10; First posted 2017-02-14 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Stomach Neoplasms
MeSH Terms: conditions — Stomach Neoplasms | interventions — HhAntag691

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- vismodegib arm (Experimental): . Vismodegib 150 mg will be administered orally once a day for 21 days as one cycle.
  Interventions: Drug: Vismodegib 150 mg

INTERVENTIONS:
Drug: Vismodegib 150 mg — Vismodegib 150 mg will be administered orally once a day for 21 days as one cycle.

SUMMARY:
There is no accepted standard therapy for patients with advanced gastric cancer who have progressed during or after second-line therapy. The role of 3rd line treatment in advanced gastric cancer has not been proven.

As a novel target of gastric cancer, SMO overexpression is chosen in this study, and the investigators plan this study to evaluate the efficacy and safety of vismodegib in gastric cancer. The doses of vismodegib are based on trials of basal cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of fully informed consent prior to any study specific procedures.
2. Patients must be ≥20 years of age.
3. Advanced gastric adenocarcinoma (including GEJ) that has progressed during or after 1st line or second-line therapy.

   * Both fluoropyrimidine and platinum agent need to be contained in the prior chemotherapies
   * Prior adjuvant or neoadjuvant therapy is counted as 1 regimen, provided that disease progression occurs within 6 months after the completion of adjuvant or neoadjuvant therapy.
   * Acceptable prior chemotherapy regimens for this protocol are chemotherapy regimens that include Immune Target agent therapy. (such as a pembrolizumab, ramucirumab etc)
4. Have the presence of measurable disease as defined by the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
5. Patients with SMO overexpression by IHC
6. Patients are willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.
7. ECOG performance status 0-1.
8. Patients must have a life expectancy ≥ 3 months from proposed first dose date.
9. Patients must have acceptable bone marrow, liver and renal function measured within 28 days prior to administration of study treatment as defined below:

   * Haemoglobin ≥9.0 g/dL (transfusion allowed)
   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   * White blood cells (WBC) > 3 x 109/L
   * Platelet count ≥100 x 109/L (transfusion allowed)
   * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) (does not include patients with Glibert's disease)
   * AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present in which case it must be ≤ 5x ULN
   * Serum creatinine ≤1.5 x institutional ULN
10. Negative urine or serum pregnancy test within 28 days of study treatment, confirmed prior to treatment on day 1. for women of childbearing potential.
11. Provision of consent for mandatory biopsy at progression (fresh frozen will be mandatory if clinically feasible)
12. Provision of archival or fresh tissue sample at baseline (fresh frozen will be mandatory if clinically feasible)

Exclusion Criteria:

Patients will be excluded from the study if they meet any of the following criteria:

1. Are currently enrolled in, or discontinued within the last 21 days from, a clinical trial involving an investigational product or non-approved use of a drug or device, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
2. Any previous treatment with Hedgehog pathway inhibitor
3. Patients with second primary cancer, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for ≤5 years.
4. HER2 positive patients (defined by HER2 3+ by immunohistochemistry or HER2 SISH +)
5. Patients unable to swallow orally administered medication.
6. Treatment with any investigational product during the last 21 days before the enrollment (or a longer period depending on the defined characteristics of the agents used).
7. Patients receiving any systemic chemotherapy, radiotherapy (except for palliative reasons), within 3 weeks from the last dose prior to study treatment (or a longer period depending on the defined characteristics of the agents used). The patient can receive a stable dose of bisphosphonates or denusomab for bone metastases, before and during the study as long as these were started at least 4 weeks prior to treatment.
8. With the exception of alopecia, any ongoing toxicities (>CTCAE grade 1) caused by previous cancer therapy.
9. Intestinal obstruction or CTCAE grade 3 or grade 4 upper GI bleeding within 4 weeks before the enrollment.
10. Resting ECG with measurable QTcB > 480 msec on 2 or more time points within a 24 hour period or family history of long QT syndrome.
11. Patients with cardiac problem as follows: Atrial fibrillation with a ventricular rate >100 bpm on ECG at rest , Symptomatic heart failure (NYHA grade II-IV), Prior or current cardiomyopathy, Severe valvular heart disease, Uncontrolled angina (Canadian Cardiovascular Society grade II-IV despite medical therapy), Acute coronary syndrome within 6 months prior to starting treatment
12. Female patients who are breast-feeding or child-bearing and Male or female patients of reproductive potential who are not employing an effective method of contraception
13. Any evidence of severe or uncontrolled systemic disease, active infection, active bleeding diatheses or renal transplant, including any patient known to have hepatitis B, hepatitis C or human immunodeficiency virus (HIV) (HBV carrier is allowed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) by RECIST 1.1 | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeeyun Lee, MD, PhD, Principal Investigator — Division of Hematology-Oncology, SMC
Locations (1):
- Samsung Medical Center, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kim R, Ji JH, Kim JH, Hong JY, Lim HY, Kang WK, Lee J, Kim ST. Safety and anti-tumor effects of vismodegib in patients with refractory advanced gastric cancer: A single-arm, phase-II trial. J Cancer. 2022 Jan 9;13(4):1097-1102. doi: 10.7150/jca.67050. eCollection 2022. PMID 35281856